CLINICAL TRIAL: NCT04444544
Title: Changes of Health-related Quality of Life 6 Months After High-risk Oncological Upper Gastrointestinal and Hepatobiliary Surgery: a Single-centre Prospective Observational Study (ChangeQol Study)
Brief Title: Quality of Life and High-Risk Abdominal Cancer Surgery
Acronym: ChangeQoL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Julien Maillard, Principal Investigator, University Hospital, Geneva
Other Study IDs: 2020-00536
Record Dates: First submitted 2020-03-12; First posted 2020-06-23 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Quality of Life; Surgery; Cancer; Frailty
Keywords: Quality of Life; Surgery; Regret
MeSH Terms: conditions — Neoplasms; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: High Risk Abdominal Surgery — Pancreatectomy, Esophagectomy, Gastrectomy and Hepatectomy

SUMMARY:
The investigators plan to measure the changes of health-related quality of life (HRQoL) at 6 months and 12 months after the following high-risk oncological abdominal surgery: gastrectomy, esophagectomy, pancreatectomy and hepatectomy. The investigators will measure the HRQoL using the validated EORTC QLQ-C30 questionnaire before and at 6 months and 12 month after the surgery. The investigators will identify phenotypes of HRQoL changes (improvement, stability and deterioration) at 6 months and 12 months after surgery.

The second aim is to assess the regret of the patient at 6 months and 12 months regarding his/her decision to undergo surgery. The investigators will also assess the regret of the next of kin at 6 months regarding the decision to undergo surgery.

This descriptive, prospective, observational, single-centre cohort study aims to: identify phenotypes of HRQoL changes after abdominal surgical oncology (improvement, stability and deterioration); assess the regret of patients regarding their decision to undergo surgical oncology at 6 months and 12 months; assess the regret of the next of kin regarding the decision of the patient to undergo surgical oncology at 6 months and 12 months. The investigators will include patients scheduled for the following elective abdominal cancer surgery: gastrectomy; esophagectomy; pancreas resection and hepatectomy. The investigators will assess HRQoL using the validated EORTC QLQ-C30 Summary Score before and 6 months and 12 months after surgery. The cut-offs for the three phenotypes of HRQoL changes will be defined using the minimal clinically important difference (MCID) of 10 points. The investigators will assess regret using the Decision Regret Scale (DRS) at 6 months and 12 months after surgery.

The expected results are: The investigators can identify phenotypes of HRQoL changes after surgical oncology using the EORTC QLQ-C30 Summary Score; the investigators will describe the distribution of these phenotypes and will find an association with the pre-existing frailty. The investigators can describe the extent of the regret of the patient and of the next of kin at 6 months using the DRS. The investigators will observe an association between the DRS score at 6 months and the HRQoL Summary Score change. The investigators will not observe a relationship between the DRS score of patients and next-of-kins.

ELIGIBILITY:
Inclusion Criteria:

- Adult patients (>18 years) scheduled for the following elective abdominal cancer surgery known for high one-year mortality4: gastrectomy; esophagectomy; pancreas resection and hepatectomy

Exclusion Criteria:

* Patients with inoperable tumours; i.e. some patients will be excluded at the time of surgery if unexpected advanced tumour staging is confirmed intraoperatively (e.g. peritoneal carcinomatosis or any other diagnosis without therapy).
* Hepatectomy for metastasectomy
* Mentally impaired patients (known diagnosis)
* Psychotic diagnoses (i.e. schizophrenia)
* Dementia (mini mental score (MMSE) < 18)
* Incapacity to understand the information sheet
* Blindness (unable to perform the visual part of the mini-mental state examination)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elective patients scheduled for high-risk abdominal cancer surgery
Sampling Method: Probability Sample
Enrollment: 295 (Estimated)
Dates: Start 2020-09-05 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Health-related Quality of Life | 6 months after surgery
  EORTC-QLQ C30. Minimum 0, Maximum 100

SECONDARY OUTCOMES:
Regret | 6 and 12 months after surgery
  Decision Regret Scale. Minimum 0, Maximum 100
Health-related Quality of Life | 12 months after surgery
  EORTC-QLQ C30. Minimum 0, Maximum 100

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of Geneva, Geneva, Switzerland

REFERENCES:
- [Derived] Maillard J, Elia N, Ris F, Courvoisier DS, Zekry D, Labidi Galy I, Toso C, Monig S, Zaccaria I, Walder B. Changes of health-related quality of life 6 months after high-risk oncological upper gastrointestinal and hepatobiliary surgery: a single-centre prospective observational study (ChangeQol Study). BMJ Open. 2023 Feb 22;13(2):e065902. doi: 10.1136/bmjopen-2022-065902. PMID 36813502